CLINICAL TRIAL: NCT04077853
Title: Efficacy of 17-Hydroxyprogesterone Caproate in Expectantly Managed Early-onset Preeclampsia: A Randomized Controlled Study
Brief Title: Progesterone in Expectantly Managed Early-onset Preeclampsia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PPET
Record Dates: First submitted 2019-09-01; First posted 2019-09-04 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Preeclampsia
MeSH Terms: conditions — Pre-Eclampsia | interventions — 17 alpha-Hydroxyprogesterone Caproate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): women will be given 17-OHPC 250 mg intra-muscular at admission and every 7 days thereafter in addition to other conservative measures of early-onset PE
  Interventions: Drug: 17 Hydroxyprogesterone Capronate
- control group (No Intervention): No intervention will be given apart from the usual conservative measures of early-onset PE

INTERVENTIONS:
Drug: 17 Hydroxyprogesterone Capronate — Intramuscular injection 250 mg
  Arms: study group

SUMMARY:
Preeclampsia is a disorder of widespread vascular endothelial malfunction and vasospasm that occurs after 20 weeks' gestation and can present as late as 4-6 weeks postpartum

DETAILED DESCRIPTION:
Currently there is no effective treatment for early-onset preeclampsia except for early delivery of the fetus along with the placenta. Progesterone supplementation in the form of 17-alpha-hydroxyprogesterone caproate (17-OHPC) is currently used obstetrically to prevent recurrent preterm birth in patients with pregnancies not complicated by preeclampsia. Previous studies reported that patients with severe PE had significantly lower serum progesterone concentrations than gestational age- and race-matched non-preeclamptics. Moreover, supplementation of placental ischemic rats with 17-OHPC decreased blood pressure, inflammatory cytokines, and ET-1 within 24 hours of treatment

ELIGIBILITY:
Inclusion Criteria:

* Gestational age between 20+0 and 33+6 weeks.
* Singleton pregnancy.
* Willing to participate in the study and sign the informed consent.

Exclusion Criteria:

* Maternal compromise requiring emergent delivery (ongoing placental abruption, DIC, pulmonary edema).
* Fetal compromise requiring emergent delivery (fetal bradycardia, recurrent late fetal heart rate decelerations).
* Platelet count < 100,000/microliter (thrombocytopenia) with evidence of HELLP syndrome;
* Persistently abnormal hepatic enzyme concentrations (twice or more upper normal values);
* Severe fetal growth restriction (ultrasound-estimated fetal weight less than fifth percentile);
* Severe Oligohydramnios (AFI < 5cm)
* Reversal of end diastolic flow(REDF) in umbilical artery Doppler testing;
* Eclampsia;
* Nonreassuring fetal status during daily testing (biophysical profile <4/10 and/or recurrent variable or late decelerations);
* Intrauterine fetal death.
* Patient is unable or unwilling to give consent.
* Patients currently using progesterone for other indications.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-12-15 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2022-01-15 (Actual)

PRIMARY OUTCOMES:
The mean difference between blood pressure measurements in both groups | one month
  blood pressure measured by mercury sphygmomanometer

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Abbas, Assiut, Cairo Governorate, Egypt